CLINICAL TRIAL: NCT04671537
Title: Effectiveness of Preloading Before Beach Chair Position on Patients Undergoing Arthroscopic Shoulder Surgery: Randomized Controlled Trial
Brief Title: The Effects of Preloading Before Beach Chair Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/166711
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Shoulder Injuries; Anesthesia; Hemodynamic Instability
Keywords: beach chair position; arthroscopic shoulder surgery; preloading; hemodynamic stability; postoperative nausea and vomiting
MeSH Terms: conditions — Shoulder Injuries; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Study group - Control group
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (preloading with crystalloid fluid - isotonic solution) (Experimental): Preloading with crystalloid fluid (isotonic solution) at 10 ml/kg of ideal body weight
  Interventions: Drug: Preloading with crystalloid fluid
- Control group (not preloading) (No Intervention): no preloading

INTERVENTIONS:
Drug: Preloading with crystalloid fluid — crystalloid fluid at 10 ml/kg of ideal body weight was administered intravenously in 30 min before the BCP for patients
  Arms: Study group (preloading with crystalloid fluid - isotonic solution)

SUMMARY:
The main objective of this study is whether preloading before positioning would be effective for less hemodynamic instability. The study also analyzes that patients with preloading will decrease postoperative nausea and vomiting, better surgical satisfaction and shortened the duration of surgery and anesthesia.

DETAILED DESCRIPTION:
Keeping patients in normovolemic state and hemodynamically stable in anesthesia and intensive care practice are important goals of anesthesiologist. It is known that hypotension that develops after taking patients to the beach chair position has a negative effect on cerebral oxygenation. Aggressive fluid regimes using to prevent hypotension can cause glycocalyx damage, edema and organ dysfunction. Also hypertension seconday to vasopressor therapy can cause bleeding at the surgical site and impaired surgical visualization during the arthroscopic shoulder surgery.

In the literature, there are studies examine whether the hypotension is the result of decreased cardiac output or decreased systemic resistance and what should be the optimal treatment , but as far as investigators know, there is no study about effects of preloading before the beach chair position on hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective arthroscopic shoulder surgery in the BCP,
* age older than 18 years and younger than 65 years,
* the American Society of Anesthesiologist (ASA) physical status of I or II,
* accepting the study protocol.

Exclusion Criteria:

* preoperative arrhythmia,
* significant heart failure
* valvular heart disease,
* preexisting cerebrovascular disease,
* deciding to switch to open surgery,
* vasopressor infusion during the surgery,
* using angiotensin converting enzyme inhibitors (ACEI) orangiotensin receptor blockers (ARB) as antihypertensive medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | during surgery (spesicific time intervals (after induction - after BCP position - 0th min - 5th min - 10th min- 30th min- 60th min)
  (mmHg)
Cardiac output | during surgery (spesicific time intervals (after induction - after BCP position - 0th min - 5th min - 10th min- 30th min- 60th min)
  (L/min)
Stroke volume variation | during surgery (spesicific time intervals (after induction - after BCP position - 0th min - 5th min - 10th min- 30th min- 60th min)
  (%) data obtained from arterial contour analysis
Heart rate | during surgery (spesicific time intervals (after induction - after BCP position - 0th min - 5th min - 10th min- 30th min- 60th min)
  bpm

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | in postoperative first day
  PONV rates
Surgical satisfaction rate | in postoperative first day
  Surgical satisfaction scale (0-10, 0 lowest score, 10 highest score) (score)
The duration of anesthesia and surgery | during surgery
  The duration of anesthesia and surgery (min)
Ephedrine usage | during surgery
  total ephedrine dose (mg) used during surgery
Total amount of crystalloid and colloid | during surgery
  Total amount of crystalloid and colloid (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Huru Ceren Gokduman, MD, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology; Elif Aygun, MD, Study Chair — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology; Nur Canbolat, MD, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology; Mert Canbaz, MD, Study Director — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology; Ali Ersen, MD, Study Chair — Istanbul Unıversity, Istanbul Faculty of Medicine Traumatology and Orthopedics; Mehmet Buget, MD, Study Chair — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology
Locations (1):
- Istanbul Unıversity, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsen SL, Lyngeraa TS, Maschmann CP, Van Lieshout JJ, Pott FC. Cardiovascular consequence of reclining vs. sitting beach-chair body position for induction of anesthesia. Front Physiol. 2014 May 19;5:187. doi: 10.3389/fphys.2014.00187. eCollection 2014. PMID 24904427
- [Background] Woodcock TE, Woodcock TM. Revised Starling equation and the glycocalyx model of transvascular fluid exchange: an improved paradigm for prescribing intravenous fluid therapy. Br J Anaesth. 2012 Mar;108(3):384-94. doi: 10.1093/bja/aer515. Epub 2012 Jan 29. PMID 22290457
- [Background] Chamos C, Vele L, Hamilton M, Cecconi M. Less invasive methods of advanced hemodynamic monitoring: principles, devices, and their role in the perioperative hemodynamic optimization. Perioper Med (Lond). 2013 Sep 17;2(1):19. doi: 10.1186/2047-0525-2-19. PMID 24472443